CLINICAL TRIAL: NCT06999499
Title: Development of Artificial Intelligence Algorithms to Help Detect Potential Melanomas, Using Images From the VECTRA 3D Whole Body 360 Imaging System, a 3D Whole-body Skin Scanner.
Brief Title: Development of an Aid to Melanoma Detection Using Artificial Intelligence Algorithms Based on Images From the VECTRA 3D System.
Acronym: SELF DETECT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RCAPHM20_0438; 2025-A01109-40 (Other: IDRCB)
Record Dates: First submitted 2025-05-20; First posted 2025-05-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Naevi
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scanner of the whole body sing the VECTRA 3D (Experimental): Whole body image acquisition using the VECTRA 3D Whole Body 360 Imaging System to detect potential melanoma
  Interventions: Other: Scanner of the whole body using the VECTRA 3D

INTERVENTIONS:
Other: Scanner of the whole body using the VECTRA 3D — Whole body image acquisition using the VECTRA 3D Whole Body 360 Imaging System to detect potential melanoma

SUMMARY:
The background to this research is that frequent medical screening of the general population for melanoma is not feasible. The real challenge of this project is to develop an automatic process for detecting any potential melanoma. To this end, the project aims to design an algorithm to build a novel diagnostic aid that makes use of the similarity and disparity of pigmented lesions in the same patient. To achieve this, we need to obtain and structure a large database of images grouping all pigmented lesions per patient according to their similarities as perceived by dermatologists.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and over
* Patient with more than 15 nevi (moles) of various phototypes (I to III)
* Patient who has received information about the study and has not expressed any opposition
* Patient who is a beneficiary or entitled person under a social security scheme

Exclusion Criteria:

* Patients with phototype V
* Patients with chronic inflammatory skin diseases
* Claustrophobic patients
* Patients who are bedridden or handicapped
* Patients who are excluded from another research protocol at the time of collection of the non-objection.
* Patients covered by articles L1121-5 to 1121-8 of the French Public Health Code (minors, adults under guardianship or trusteeship, patients deprived of their liberty, pregnant or breast-feeding women),
* Any other reason which, in the investigator's opinion, could interfere with the evaluation of the research objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
development and validation of algorithms to identify lesions clinically suspected of being melanoma by a dermatologist (potentially malignant and/or ugly duckling). | from enrollement to until 6 month
  Comparison of the results given by the analysis of the images by 3 dermatologists or by the software. Estimation of sensitivity and specificity thresholds of at least 93% (accuracy level 5%).

SECONDARY OUTCOMES:
concordance rate for malignant annotations | From enrollement to 6 month after
  concordance between the malignant yes-no annotations of each of the three dermatologists (2 to 2) will be tested.
concordance rate for ugly duckling | From enrollement to 6 month after
  concordance between the ugly duckling yes-no annotations of each of the three dermatologists (2 to 2) will be tested.
calculation of the proportion of melanomas confirmed by anatomopathology | From enrollement to 6 month after
  For each lesion identified as malignant or ugly duckling by the gold standard and removed for histological analysis: calculation of the proportion of melanomas confirmed by pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Conception, Marseille, France